CLINICAL TRIAL: NCT01314027
Title: Adjuvant Gemcitabine Versus NEOadjuvant Gemcitabine/Oxaliplatin Plus Adjuvant Gemcitabine in Resectable PAncreatic Cancer: a Randomized Multicenter Phase III Study (NEOPAC Study)
Brief Title: Adjuvant Versus Neoadjuvant Plus Adjuvant Chemotherapy in Resectable Pancreatic Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low recruitment
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEOPAC
Record Dates: First submitted 2010-09-29; First posted 2011-03-14 (Estimated); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Neoadjuvant Therapy; Gemcitabine; Oxaliplatin; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- neoadjuvant + adjuvant chemotherapy (Experimental): neoadjuvant chemotherapy is based on gemcitabine/oxaliplatin adjuvant therapy is based on gemcitabine
  Interventions: Drug: Neoadjuvant Chemotherapy with gemcitabine/oxaliplatin
- adjuvant chemotherapy (Active Comparator): adjuvant therapy is based on gemcitabine
  Interventions: Drug: adjuvant chemotherapy with gemcitabine

INTERVENTIONS:
Drug: Neoadjuvant Chemotherapy with gemcitabine/oxaliplatin — Patients with resectable cytologically proven adenocarinoma of the pancreatic head are randomized to arm A or B.
  Patients randomized to arm A receive an 8-week neoadjuvant chemotherapy with gemcitabine/oxaliplatin. Thereafter, surgery is performed if the restaging does not reveal a contraindication. Finally, all patients receive adjuvant gemcitabine for six months.
  Other Names: gemcitabine; eloxatin
  Arms: neoadjuvant + adjuvant chemotherapy
Drug: adjuvant chemotherapy with gemcitabine — Patients randomized to arm B undergo surgery and receive the same adjuvant treatment as in arm A.
  Arms: adjuvant chemotherapy

SUMMARY:
The outcome of patients with resected pancreatic cancer has significantly been improved by adjuvant chemotherapy. However, a large proportion of patients cannot receive adjuvant chemotherapy due to surgical complications. Neoadjuvant chemotherapy has been shown to be safe and effective and can be applied to all patients. This study should test neoadjuvant chemotherapy in a randomized manner.

Patients with resectable cytologically proven adenocarinoma of the pancreatic head are randomized to arm A or B.

Patients randomized to arm A receive an 8-week neoadjuvant chemotherapy with gemcitabine/oxaliplatin followed by surgery. Thereafter, all patients receive adjuvant gemcitabine for six months.

Patients randomized to arm B undergo surgery and receive the same adjuvant treatment as in arm A.

The primary study-endpoint is the recurrence-free survival. Tumor recurrence are determined by computed tomography in a defined protocol.

* Trial with medicinal product

DETAILED DESCRIPTION:
Due to the improvement in the recurrence-free and overall survival by adjuvant chemotherapy, surgery followed by adjuvant chemotherapy is currently considered the standard treatment for resectable pancreatic cancer. However, a significant proportion (>25%) of patients cannot receive adjuvant treatment due to the morbidity of pancreas surgery. Neoadjuvant (preoperative) chemotherapy appears particularly attractive since it can be applied to all patients and has resulted in a significant histological tumor response with a median survival superior to adjuvant chemotherapy in a recent prospective phase II trial.

The aim of this study is to determine the role of neoadjuvant chemotherapy in patients with resectable pancreatic cancer.Eligible patients are randomized to:

arm A: neoadjuvant chemotherapy + resection + adjuvant chemotherapy arm B: resection + adjuvant chemotherapy Neoadjuvant chemotherapy consists of gemcitabine (1000mg/m2) and oxaliplatin (100mg/m2) on days 1, 15, 29 and 43, while adjuvant chemotherapy is based on gemcitabine 1000mg/m2 for 6 months.

If the restaging protocol excludes distant metastases, a diagnostic laparoscopy is performed, followed by a Whipple operation in the absence of distant metastases.

The primary study end-point is the recurrence-free survival after study inclusion, and this is defined by the interval between the date of written informed consent until recurrence. Secondary end-points are the overall survival and the surgical complication rate. Interim analyses are performed after the inclusion of 100 and 200 patients without interrupting patient accrual. An independent data monitoring committee will review the results of each interim analysis and will decide about the study cessation or continuation.

Patients will be followed-up according to the protocol below in order to assess tumor recurrence.

Quality of life will be assessed by the QLQ-30 questionnaire of the EORTC at study entry, after neoadjuvant chemotherapy, start and end of the adjuvant chemotherapy and at each follow-up study visit. Representative histological samples are reviewed and stored by the reference pathologist at the University Hospital of Zurich. These samples will also be used to determine the histological response and extent of cytopathic effects. Furthermore, the nutritional status is assessed from all patients by the prealbumin serum levels at study entry and prior to surgery. Further translational research is desired and will be individually organized by each center.

ELIGIBILITY:
Inclusion criteria:

* resectable adenocarcinoma of the pancreatic head (requiring duodeno-pancreatectomy)
* T1-3, Nx, M0 (UICC 6th version, 2002)
* infiltration of the portal vein (<180°) is not an exclusion criterion
* cytologic or histologic confirmation of adenocarcinoma
* age >18 years
* written informed consent

Exclusion criteria:

* contraindication for Whipple procedure
* an infiltration >180° of the portal vein
* abutment of the tumor to the superior mesenteric artery
* infiltration of the superior mesenteric artery or the celiac trunk
* chronic neuropathy > grade 2
* WHO performance score >2
* uncorrectable cholestasis (bilirubin > 100mmol/l despite drainage attempts for more than four weeks prior to inclusion)
* female patients in child bearing age not using adequate contraception (oral or subcutaneous contraceptives, intrauterine pessary (IUP), condoms)
* pregnant or lactating women
* mental or organic disorders which could interfere with giving informed consent or receiving treatments
* Second malignancy diagnosed within the past 5 years, except non-melanomatous skin cancer or non-invasive cervical cancer
* percutaneous biopsy of the primary tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-09; Primary Completion 2018-12 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 9 months after inclusion
  by computed tomography

SECONDARY OUTCOMES:
Progression-free survival | 12, 15, 21, 27, 33, 39, ... months after inclusion
  by computer tomography
histological response | Pancreatic resection
  Histology
overall survival | 1, 3 and 5 years after inclusion
complication rates after surgery | 60 days postoperative
feasibility of adjuvant chemotherapy | within 8 postoperative weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Alain Clavien, MD, PhD, Study Director — UniversitaetsSpital Zuerich
Locations (5):
- University Hospital of Gent, Ghent, Belgium
- France (2):
  - University Hospital of Marseille, Marseille
  - University Hospital of Strasbourg, Strasbourg
- University Hospital Mainz, Mainz, Germany
- University Hospital of Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Heinrich S, Pestalozzi B, Lesurtel M, Berrevoet F, Laurent S, Delpero JR, Raoul JL, Bachellier P, Dufour P, Moehler M, Weber A, Lang H, Rogiers X, Clavien PA. Adjuvant gemcitabine versus NEOadjuvant gemcitabine/oxaliplatin plus adjuvant gemcitabine in resectable pancreatic cancer: a randomized multicenter phase III study (NEOPAC study). BMC Cancer. 2011 Aug 10;11:346. doi: 10.1186/1471-2407-11-346. PMID 21831266